CLINICAL TRIAL: NCT05248542
Title: The Effects of Virtual Reality/ Augmented Reality Usage on Oral Care Knowledge in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KMUHIRB-SV(II)-20200062
Record Dates: First submitted 2021-12-30; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2021-12

CONDITIONS: Virtual Reality; Oral Care; Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality group (Experimental): Each participant in the experimental group received a 30 minutes of individualized VR-based simulation education in a dedicated oral skills training room.
  Interventions: Other: Virtual Reality Usage on Oral Care Knowledge
- Control group (No Intervention): The control group only received repeated questionnaires and did not receive any education about geriatric oral hygiene.

INTERVENTIONS:
Other: Virtual Reality Usage on Oral Care Knowledge — Virtual Reality Usage on Oral Care Knowledge about independent older adults
  Arms: Virtual Reality group

SUMMARY:
The aim of this study was to investigate the effects of virtual reality usage on oral care knowledge in nursing students. The participants were randomly assigned to virtual-reality experimental and control groups. The students in experimental group received a 30 minutes virtual reality (VR) training for elderly oral health care at the second week and the fourth week after the first time survey. All students self-administrated questionnaire three times at first date of consent form signed, immediately after each of the intervention for period of two weeks. Linear regression in generalized estimating equations (GEE) compare the differences between both groups.

DETAILED DESCRIPTION:
A total of 50 first-year to third-year undergraduate nursing students were included from the Department of Nursing, Kaohsiung Medical University, Taiwan. The students were randomly assigned divided at random into two groups, control (n = 25) and experimental (n = 25).

ELIGIBILITY:
Inclusion Criteria:

1. undergraduate freshman, sophomore, and junior nursing students
2. those volunteered to participate in this study

Exclusion Criteria:

1. students with known negative effects of using VR devices, such as nausea, vomiting, etc.
2. those under 20 years of age who had not obtained the consent of a legal representative to participate in this study.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Knowledge of geriatric oral hygiene scale | through study completion, an average of 4 weeks
  There were 10 items to evaluate the participants' knowledge of the geriatric oral hygiene scale Each item had three response options: true, false, and unknown. The total score ranged from 0 to 10 and a higher score indicated a higher level of knowledge of geriatric oral hygiene.
Attitudes of geriatric oral hygiene scale | through study completion, an average of 4 weeks
  The attitudes of geriatric oral hygiene scale included seven items. Each item was scored on a five-point Likert-type scale ranging from 1 (strongly disagree) to 5 (strongly agree). The total score ranged from 5 to 35 and a higher score indicated a positive attitude toward geriatric oral hygiene.
Self-efficacy of geriatric oral hygiene scale | through study completion, an average of 4 weeks
  The self-efficacy of geriatric oral hygiene scale included ten items. Each item was scored on a five-point Likert-type scale ranging from 1 (strongly disagree) to 5 (strongly agree) and the higher score was for a higher level of self-efficacy of geriatric oral hygiene, vise versa. The total score ranged from 5 to 50.
Behavioral intention of geriatric oral hygiene scale | through study completion, an average of 4 weeks
  The behavioral intention scale of the geriatric oral hygiene included ten items. Each item was scored on a five-point Likert-type scale ranging from 1 (strongly disagree) to 5 (strongly agree), with a higher score indicated a higher level of the behavioral intention of geriatric oral hygiene. The total score ranged from 5 to 50.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Chao Lin, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin PC, Wung SF, Lin PC, Lin YC, Lin CY, Huang HL. Virtual reality-based simulation learning on geriatric oral health care for nursing students: a pilot study. BMC Oral Health. 2024 May 28;24(1):627. doi: 10.1186/s12903-024-04249-y. PMID 38807116